CLINICAL TRIAL: NCT02260219
Title: Comparative Study of the Safety and Efficacy of the Ahmed Glaucoma Valve Drainage Device, Model M4 (High Density Porous Polyethylene) and the Model S2 (Polypropylene) in Patients With Neovascular Glaucoma
Brief Title: Comparative Study, Safety and Efficacy, Ahmed Glaucoma Drainage Device, Model M4 Model S2 in Neovascular Glaucoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-12-01
Record Dates: First submitted 2014-07-17; First posted 2014-10-09 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Neovascular Glaucoma
Keywords: Ahmed implant; Neovascular Glaucoma; Intraocular pressure
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S2 (Active Comparator): Surgically Implant an Ahmed Glaucoma Drainage Device Model S2 in Neovascular Glaucoma Patients and evaluate the IOP evolution, complications and need for medication to control IOP
  Interventions: Procedure: Surgical Implant of Ahmed Glaucoma Drainage Device, model M4 and S2
- M4 (Active Comparator): Surgically Implant an Ahmed Glaucoma Drainage Device Model M4 in Neovascular Glaucoma Patients and evaluate the IOP evolution, complications and need for medication to control IOP
  Interventions: Procedure: Surgical Implant of Ahmed Glaucoma Drainage Device, model M4 and S2

INTERVENTIONS:
Procedure: Surgical Implant of Ahmed Glaucoma Drainage Device, model M4 and S2 — Surgically Implant an Ahmed Glaucoma Drainage Device Models S2 and M4, evaluare IOP evolution, complications and need for medication to control IOP

SUMMARY:
Objective: Prospectively evaluate the safety and efficacy of the Ahmed Glaucoma Drainage Device, model M4 compared with the model S2.

Method: Mexican patients with Neovascular Glaucoma will be randomly included for each group (M4 and S2). They will be operated using conventional techniques and creating a sub-episcleral tunnel to place the valve's tube in the anterior chamber. They will be monitoring for one year and the results will be evaluated with respect to a postoperative reduction in pressure, changes in visual acuity, the need for drugs and complications, in addition to the demographic characteristics of each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Neovascular glaucoma
* High IOP despite topical treatment

Exclusion Criteria:

* Pregnant women
* Mental disorders
* Previous glaucoma surgery
* Patients older than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse effects | 1 year

SECONDARY OUTCOMES:
Intraocular pressure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Felix Gil-Carrasco, MD, Study Director — 52 55 10841400